CLINICAL TRIAL: NCT03174015
Title: Sanitation Demand Creation in Peri-Urban Slums of Lusaka, Zambia
Acronym: SanDem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Robert Aunger, Associate Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QA_840
Record Dates: First submitted 2017-02-22; First posted 2017-06-02 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Diarrhea
Keywords: Sanitation; Demand; Peri-urban; Behavior Change; Lusaka; Zambia
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: A random sample of plots will be selected in Bauleni Compound and invited to participate. Intervention allocation will also be randomized, with approximately equal numbers of plots allocated to the intervention and control arms. Within the chosen plots, resident landlord households will receive the intervention and resident landlord households and one randomly selected tenant household will be chosen for data collection for both intervention and control plots.
Who Masked: Outcomes Assessor
Masking Description: The study will be partially single blinded. Participants and investigators cannot be masked to the intervention but outcome assessors will not know where the intervention has taken place and will be given only minimal information to enable assessment of intervention exposure at the end of the survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Landlords on selected plots will receive the "Bauleni Secret" intervention. Landlords and selected tenants will be surveyed in baseline/end-line data collection.
  Interventions: Behavioral: Bauleni Secret
- Control (No Intervention): Landlords and selected tenants will be surveyed in baseline/end-line data collection only.

INTERVENTIONS:
Behavioral: Bauleni Secret — The intervention will invite enrolled landlords to a series of meetings in which various mechanisms will be used, each designed to increase their likelihood of improving the toilet(s) on their plot. These meetings will be the main vehicle for a status-building campaign associated with increasing wealth by improving plot sanitation, understanding tenants' implicit demand, understanding the processes by which toilets can be improved, and a competition rewarding landlords that make the greatest improvements to the improvement of their toilet(s).
  Arms: Intervention

SUMMARY:
This intervention will experimentally test the hypothesis that sanitation can be improved in a peri-urban setting using state-of-the-art behaviour change communications.

Formative research indicated that landlords are the effective decision-makers about investments in sanitation on their plots (which can include a number of tenant households as well). Landlords will therefore be the primary targets of the intervention. The study will take the form of a randomized controlled trial of the intervention evaluated at the plot level. The intervention will invite enrolled landlords to a series of meetings in which various mechanisms will be used, each designed to increase their likelihood of improving the toilet(s) on their plot. These meetings will be the main vehicle for a status-building campaign associated with increasing wealth by improving plot sanitation, understanding tenants' implicit demand, understanding the processes by which toilets can be improved, and a competition rewarding landlords that make the greatest improvements to the improvement of their toilet(s). The desired improvements will be measured via multiple primary outcomes that measure aspects of changes to hardware and software components, including indicators of hygienic quality, psychological desirability, accessibility, and ecological sustainability. This is because the investigators argue that, to have a significant impact on population-level diarrheal disease indicators, any sanitation solution must be:

* effective at reducing exposure to pathogens (i.e., hygienic),
* desirable (i.e., seen as valuable or humane), and
* accessible (i.e., no one excluded), so that it can be used by all
* for a reasonably long time (i.e., sustainable)

ELIGIBILITY:
Plots will be selected for inclusion in the study based on meeting the inclusion criteria. The intervention will be delivered to the landlord on each plot assigned to the intervention arm.

Intervention Inclusion Criteria:

* Plot located in Bauleni compound
* Adult landlord (age 18 or higher) resides on plot

Intervention Exclusion Criteria:

* None

Data will be collected from the landlord and one randomly selected tenant from all eligible adult tenants on each plot.

Data Collection Inclusion Criteria:

* Adult landlord or tenant (age 18 or higher) resides on selected plot most of the time

Data Collection Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Having a hole-cover or water-sealed pan | 5 months after intervention begins
  Reduces spread of pathogens by creating barrier between containment and above-ground environment
Having a latrine door that locks from the inside | 5 months after intervention begins
  Provide safety and privacy for toilet users
Having a latrine door that locks from the outside | 5 months after intervention begins
  Exclude those not living on the plot from the toilet
Having a rotational cleaning system in place | 5 months after intervention begins
  To maintain hygienic condition of the toilet interface

SECONDARY OUTCOMES:
Willingness to pay | 5 months after intervention begins
  Change in landlord stated willingness to pay for toilet improvements
Attitudes towards sanitation | 5 months after intervention begins
  Scales measuring landlord attitudes towards the importance of sanitation
Financial preparation for toilet improvement | 5 months after intervention begins
  Landlords report saving money, either individually or by participating in a rotating savings scheme, for toilet improvement
Partial construction progress towards toilet improvement | 5 months after intervention begins
  Landlords have either amassed raw materials on the plot (concrete blocks, wood, etc.) for toilet improvement or new construction/upgrading of toilet began (hole dug for new toilet, new slab poured for flushing toilet, etc.)
Peri-urban Healthy Toilet Index | 5 months after intervention begins
  A theory-based comprehensive index of on-site peri-urban sanitation status including hygienicity, accessibility, desirability, and sustainability of sanitation systems
Cleaning rota initiated | 5 months after intervention begins
  Landlord reports taking any action directed at establishing a rotational cleaning system (e.g., holding a plot meeting explicitly for this purpose, posting a written rota, or otherwise tangibly indicating rota responsibilities)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Aunger, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Roma Chilengi, MD, Principal Investigator — Center for Infectious Disease Research in Zambia; Valerie Curtis, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Bauleni Compound, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available with consent from the principal investigators. The study will collect only basic demographic information on individuals along with knowledge/attitudes/preferences data, so there will be little to identify individuals from the shared IPD and little that is very sensitive.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from approximately June 2018 for at least 5 year on study website.
Access Criteria: Data will be accessible with consent from study PIs per submitted proposals and protocols.
URL: http://www.shareresearch.org/project/san-dem

REFERENCES:
- [Derived] Tidwell JB, Chipungu J, Bosomprah S, Aunger R, Curtis V, Chilengi R. Effect of a behaviour change intervention on the quality of peri-urban sanitation in Lusaka, Zambia: a randomised controlled trial. Lancet Planet Health. 2019 Apr;3(4):e187-e196. doi: 10.1016/S2542-5196(19)30036-1. PMID 31029230
- See also: Study website — http://www.shareresearch.org/project/san-dem